CLINICAL TRIAL: NCT01296061
Title: Effect of Immunosuppressive Medication Use on Patient Outcomes Following Kidney Transplantation Failure
Brief Title: Kidney Transplant Failure
Status: Terminated | Type: Observational
Why Stopped: Funding ended.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); St. Paul's Hospital, Canada (Other); Vancouver General Hospital (Other); Kingston Health Sciences Centre (Other); University of Saskatchewan (Other); University of Calgary (Other); University of Manitoba (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); St. Joseph's Healthcare Hamilton (Other); London Health Sciences Centre (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Maisonneuve-Rosemont Hospital (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); CHU de Quebec-Universite Laval (Other); University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: CIHR FRN MOP-102732
Record Dates: First submitted 2011-02-08; First posted 2011-02-15 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Acute Graft Rejection; Renal Failure Chronic Requiring Dialysis
Keywords: Dialysis; Renal Transplantation; Failure of allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Class I and II HLA antibodies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Failed Kidney Transplant: Adults ≥ 18 years, initiating chronic dialysis

SUMMARY:
Primary Hypotheses:

1. Among patients who retain the failed kidney transplant, those who continue immunosuppressant medication will have more deaths than patients who discontinue these drugs
2. Among patients who retain the failed kidney transplant, those who continue immunosuppressant medication will have more hospitalizations for sepsis than patients who discontinue these drugs
3. Among patients who retain the failed kidney transplant, those who continue immunosuppressant medication will have fewer rejection events than patients who discontinue these drugs

Secondary Hypotheses:

1. Patients who undergo elective nephrectomy (to remove the failed kidney transplant) will have fewer deaths than those who retain the failed kidney transplant
2. Patients who undergo elective nephrectomy (to remove the failed kidney transplant) will have fewer hospitalizations for sepsis than those who retain the failed kidney transplant
3. Among patients who retain the failed kidney transplant, those who continue immunosuppressant medication will have lower levels of allosensitization (anti-HLA antibodies) than those who discontinue these drugs
4. Patients who undergo elective nephrectomy will have higher levels of allosensitization (anti-HLA antibodies) than patients who retain the failed kidney transplant

DETAILED DESCRIPTION:
Transplantation is the best treatment for patients with end stage kidney disease.1 However, despite the development of powerful immunosuppressant medications, transplantation still does not provide most patients with lifelong freedom from dialysis. The half-life (time to 50% failure) of a deceased donor kidney transplant is only 10.5 years.4, 5 As the number of prevalent patients who received a transplant more than a decade ago increases, the number of patients with failing transplants who must either return to dialysis or undergo repeat transplantation is also rapidly increasing.6 Repeat transplantation is clearly the best option for these patients.8 However, in Canada, only 10% of patients with first transplant failure will receive a second transplant.9 Consequently transplant failure is now the fifth leading individual cause of dialysis initiation in Canada.6, 10 Survival after transplant failure is very poor, with 40% mortality in the first 5 years after initiation of dialysis.9, 11, 12 In comparison, the 5 year mortality of de novo incident dialysis patients, including those who are not even transplant candidates, is 50%, 6, 10while that of first transplant recipients is < 10%.6, 10 However, the unique characteristics of the transplant failure population limit the validity of such comparisons with other chronic kidney disease patients. Transplant failure patients were initially selected to undergo transplantation because of their favorable age and health status, and thus differ from unselected de novo incident dialysis patients. Similarly, unlike first time transplant recipients, transplant failure patients already have prolonged exposure to immunosuppressant medications that can increase the risk of cardiovascular disease, cancer and metabolic bone disease. Notwithstanding these issues, we and others have published a number of studies documenting the poor outcomes, and stressing the need for prospective studies in this unique subset of chronic kidney disease patients.9, 12-16 To date, no study has systematically examined this patient population and basic questions about how to manage the failed kidney allograft remain. Although there are some clear indications for emergent surgical removal of the failed allograft (nephrectomy), the elective use of nephrectomy is highly variable and poorly described.17-19 Acute immunologic injury (rejection) in the failed transplant can occur as long as the allograft remains in situ, and can cause both local and systemic symptoms. In addition, the failed allograft may promote chronic inflammation leading to malnutrition, anemia and cardiovascular disease.20, 21 No prospective studies have examined whether nephrectomy and discontinuation of immunosuppressant medications is preferable to retaining the failed allograft. If the allograft is retained, it is not known whether the risk of continued exposure to immunosuppressant medications outweighs the risk of acute rejection or chronic inflammation when these drugs are discontinued. Importantly, management of the failed allograft can impact allosensitization,22-24 a primary determinant of a patient's ability to undergo repeat transplantation.

This prospective observational study is a necessary first step in defining the optimal management strategy for this unique and growing patient population. The primary and secondary research questions will determine the association of (i) immunosuppressant drug use and (ii) elective nephrectomy with clinical outcomes including death, sepsis, and rejection. Importantly, the study will also determine the association of these exposures with allosensitization (anti-HLA antibodies). The information obtained will inform the design of future interventional studies that will definitively define how to best manage these complex patients.

ELIGIBILITY:
Inclusion Criteria:Patients ≥ 18 years, who initiate chronic dialysis treatment after failure of a first kidney transplant

Exclusion Criteria:Recipients of a multi-organ transplant (e.g. kidney- pancreas transplant), and patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years, who initiate chronic dialysis treatment after failure of a first kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2011-08; Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Death | 48 months
  Death: Death will be identified through monthly contact of study coordinators with the treating dialysis center. Date of death will be obtained from records maintained by dialysis programs. If required, the patient's treating physician may contact the next of kin to confirm the date of death.
Sepsis | 48 months
  Sepsis: Hospital discharge records will be reviewed for the most responsible diagnosis. Hospitalizations for sepsis will be identified if an infection is recorded as the primary or secondary discharge diagnosis, and confirmatory laboratory evidence of infection (i.e. positive culture or chest radiograph compatible with pneumonia) is present. In the absence of laboratory evidence of infection, documentation of clinical sign or symptoms of infection will be required (fever, shock, localizing symptoms). The source of infection (e.g. catheter related, urinary tract etc) will be documented.
Rejection of failed allograft. | 48 months
  Rejection of failed allograft: After transplant failure, rejection is rarely confirmed by a biopsy of the allograft. Rejection events will be identified by patient interview and clinical chart review during follow up visits. Rejection will be identified when both a diagnosis of rejection with compatible signs/ symptoms is documented and either an increase in immunosuppressant drugs is prescribed, or transplant nephrectomy is performed. Only rejection events diagnosed after the initiation of dialysis will be included.
Allosensitization | 48 months
  Allosensitization: Serum samples will be collected at baseline and at each study visit. Dialysis centers routinely collect serum samples for monitoring allosensitization in wait-listed transplant candidates and have established local protocols for collection, storage and shipping. Both class I and class II Anti-HLA antibodies will be appraised using FlowPRA®.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Knoll, MD, Principal Investigator — U of Ottawa, The Ottawa Hospital, OHRI; John Gill, MD, Principal Investigator — UBC, St Paul's Hospital Vancouver, BC
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada